CLINICAL TRIAL: NCT06866795
Title: A Phase 1 Open-Label, Dose-Escalation and Dose-Expansion Study Evaluating the Safety, Pharmacokinetics and Clinical Activity of Orally Administered GT-220F in Subjects With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: Phase 1 Clinical Study of GT-220F in Subjects With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Geode Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GT-220F-101
Record Dates: First submitted 2025-02-28; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: prostate cancer; metastatic prostate cancer; castration resistant prostate cancer; PTEN-loss; mCRPC; PTEN-deficient; PI3K; PI3Kbeta
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- GT-220F Dose Level 1 (Experimental): GT-220F 50mg, oral capsule, once a day
  Interventions: Drug: GT-220F capsule
- GT-220F Dose Level 2 (Experimental): GT-220F increased dose level to be determined, oral capsule, once or twice a day
  Interventions: Drug: GT-220F capsule
- GT-220F Dose Level 3 (Experimental): GT-220F increased dose level to be determined (if needed), oral capsule, once or twice a day
  Interventions: Drug: GT-220F capsule
- GT-220F Dose Level 4 (Experimental): GT-220F increased dose level to be determined (if needed), oral capsule, once or twice a day
  Interventions: Drug: GT-220F capsule
- GT-220F Dose Level 5 (Experimental): GT-220F increased dose level to be determined (if needed), oral capsule, once or twice a day
  Interventions: Drug: GT-220F capsule
- GT-220F Dose Expansion (Experimental): GT-220F recommended phase 2 dose, oral capsule, once or twice a day
  Interventions: Drug: GT-220F capsule

INTERVENTIONS:
Drug: GT-220F capsule — GT-220F capsule for oral administration
  Other Names: 9-((R)-1-((3,5-difluorophenyl)amino)ethyl)-7-((R)-3-(dimethylamino)pyrrolidine-1-carbonyl)-2-morpholino-4H-pyrido[1,2-a]pyrimidin-4-one fumarate

SUMMARY:
The goal of this clinical trial is to test GT-220F in patients with metastatic castration resistant prostate cancer and learn about the best dose required for further study. Participants will be adults with metastatic castration resistant prostate cancer. The main questions the study aims to answer are: 1) What medical problems do participants have when taking GT-220F? 2) What dose strength is best to use in further clinical trials? Participants will be asked to

* take GT-220F every day
* take medical tests every week

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥ 18 years of age. Because no dosing or adverse event data are currently available on the use of GT-220F in subjects <18 years of age, children are excluded from this study.
2. In Dose Escalation (Part 1) Only - subjects must have histologically confirmed recurrent or progressive metastatic castration resistant prostate cancer (mCRPC). In Dose Expansion (Part 2) Only - subjects must have histologicaly confirmed recurrent or progressive mCRPC with alterations in the PTEN gene (mutations or deletions) or PIK3CB gene (activating mutations or amplifications) as determined by Next-Generation Sequencing.
3. Subjects must have received at least one previous AR pathway inhibitor (enzalutamide, apalutamide, darolutamide, abiraterone acetate) for biochemically recurrent or metastatic prostate cancer.
4. Ongoing ADT with a lutenizing hormone releasing hormone agonist/antagonist or bilateral orchiectomy that results in serum testosterone < 50 ng/dL.
5. Subjects must have shown evidence of radiological and/or prostate specific antigen (PSA) progression. For PSA progression, there must be at least 2 sequential rises at a minimum of 1-week intervals. The first PSA value must be ≥ 2 ng/mL. Progression of measurable disease (RECIST 1.1 criteria) or presence of at least two new bone lesions (Prostate Cancer Working Group 3 criteria).
6. Subjects must have recovered to grade ≥ 2 or pre-treatment baseline from clinically significant toxic effects of prior therapy.
7. ECOG performance status >2
8. Subjects must have adequate organ and marrow function as defined below:

   1. absolute neutrophil count ≥ 1,500/mcL
   2. hemoglobin ≥ 9g/dL
   3. platelets ≥ 75,000/mcL
   4. total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (subjects with Gilbert syndrome are allowed if direct bilirubin within normal limits)
   5. AST(SGOT)/ALT(SGPT) ≤ 3 x institutional ULN
   6. creatinine ≤ 1.5 xULM mg/dL OR a calculated creatinine clearance ≥50mL/min.
9. Left ventricular ejection fraction at least 50% by echocardiogram or multigated acquisition scan.
10. Subjects with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, subjects should be class 2B or better.
11. Men who partner with a woman of childbearing potential must agree to use effective, dual contraceptive methods (i.e., a condom, with female partner using oral, injectable or barrier method) while on study drug and for 4 months afterward.
12. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Evidence of oncogenic mutations in PIK3CA, RAS or receptor tyrosine kinase (RTK) genes (EGFR, ALK).
2. Subjects who have had prior treatment with PI3K inhibitors with beta and/or delta isoform activity: GSK2636771, AZD 8186, idelalisib, copanlisib, duvelisib, umbralisib.
3. Subjects who have had any cancer-directed immunomodulatory or molecularly-targeted agent or monoclonal antibody within 14 days prior to initiation of study drug.
4. Subjects who have used any investigational agents within 28 days or 5 half-lives from study initiation, whichever is shorter.
5. Subjects who have increasing corticosteroid requirement or a dose >6 mg per day of dexamethasone or equivalent dose of other corticosteroids within 7 days prior to study initiation.
6. Subjects who received radiation therapy within 4 weeks prior to enrollment, unless there is surgical confirmation of recurrent disease or evidence of new enhancing recurrent disease outside of the prior radiotherapy treatment field.
7. Subjects who have had major surgery within 28 days prior to registration.
8. Subjects with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to GT-220F.
9. Subjects with known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness.
10. Subjects with any of the following within 6 months prior to initiation of study drug: uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack.
11. Pulmonary embolism within 1 month prior to initiation of study drug.
12. Unstable cardiac dysrhythmias or persistent prolongation of the QTc (Fridericia) interval to >470msec.
13. Evidence of Grade ≥ 2 intracranial hemorrhage.
14. Subjects with any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the Investigator's opinion, would make the subject inappropriate for entry into this study.
15. Subjects with uncontrolled intercurrent illness, including active or clinically unstable bacterial, viral or fungal infection requiring systemic therapy.
16. Subjects with difficulty swallowing/unable to swallow pills; malabsorption syndrome; refractory nausea and vomiting, chronic gastrointestinal (GI) disease or previous significant bowel resection with clinically significant sequelae that would preclude adequate absorption of study drug.
17. Another cancer for which they are receiving active treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | at the end of Cycle 1 (each cycle is 28 days)
  Number and severity of dose limiting toxicity during Cycle 1 of GT-220F administration during dose escalation
Maximum Tolerated Dose (MTD) | at the end of Cycle 1 (each cycle is 28 days)
  Maximum tolerated dose, determined by the occurrence of dose limiting toxicities during Cycle 1 of GT-220F administration
Recommended Phase 2 Dose | at the end of Cycle 1 (each cycle is 28 days)
  Recommended Phase 2 dose, determined by evaluation of maximum tolerated dose, dose limiting toxicities, and pharmacokinetics during Cycle 1 of GT-220F administration
Adverse Events | from date of randomization to date of progression, assessed up to 50 weeks
  Adverse events, characterized by type, frequency and relationship to the intervention (GT-220F) during administration of GT-220F and for 30 days after stopping administration of GT-220F

SECONDARY OUTCOMES:
Objective tumor response rate (ORR) | from date of randomization to date of progression, assessed up to 50 weeks
  The number of subjects achieving objective response [complete response (CR) and partial response (PR)] divided by number of subjects who initiate treatment
Duration of objective tumor response (DOR) | from date of randomization to date of progression, assessed up to 50 weeks
  The duration of objective response will be measured from the time measurement criteria are met for complete reponse or partial response (whichever is first recorded) until the first date that recurrent or progressive disease (PD) is documented
Disease control rate (DCR) | from date of randomization to date of progression, assessed up to 50 weeks
  The percentage of patients who experience complete response, partial response, or stable disease (SD)
Radiographic progression-free survival (PFS) | from date of randomization to date of progression, assessed up to 50 weeks
  Time from treatment initiation to the earlier of (1) disease progression by RECIST1.1 and/or Prostate Cancer Working Group 3 criteria or (2) death due to to any cause.
Prostate specific antigen measurements - change from baseline | from date of randomization to date of progression, assessed up to 50 weeks
  Proportion of patients achieving 30%, 50% or 90% reduction in prostate specific antigen (PSA) measurement from baseline.
Area under the curve (AUC) | 22 days from baseline
  Pharmacokinetic assessment of area under the curve (AUC) for GT-220F and GT-220F-M1 (active metabolite)
Maximum plasma concentration (Cmax) | 22 days from baseline
  Pharmacokinetic assessment of maximum plasma concentration (Cmax) for GT-220F and GT-220F-M1 (active metabolite)
Trough plasma concentration (Cmin) | 22 days from baseline
  Pharmacokinetic assessment of trough plasma concentration (Cmin) for GT-220F and GT-220F-M1 (active metabolite)
Time to maximum plasma concentration (Tmax) | 22 days from baseline
  Pharmacokinetic assessment of time to maximum plasma concentration (Tmax) for GT-220F and GT-220F-M1 (active metabolite)
Plasma half-life (T1/2) | 22 days from baseline
  Pharmacokinetic assessment of plasma half-life (T1/2) for GT-220F and GT-220F-M1 (active metabolite)
Plasma clearance (CL) | 22 days from baseline
  Pharmacokinetic assessment of plasma clearance (CL) for GT-220F and GT-220F-M1 (active metabolite)
Volume of distribution | 22 days from baseline
  Pharmacokinetic assessment of volume of distribution for GT-220F and GT-220F-M1 (active metabolite)

CONTACTS AND LOCATIONS:
Overall Officials: Alok Tewari, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: No